CLINICAL TRIAL: NCT07061613
Title: Evaluating the Efficacy and Safety of NeoThelium FT Amnion Skin Graft in the Management of Venous Leg Ulcers: A Prospective Case Series
Brief Title: Prospective Case Series Evaluating the Efficacy and Safety of NeoThelium FT for Venous Leg Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoVein
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Venous Leg Ulcer
Keywords: Chronic Wounds; Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: NeoThelium FT in addition to Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoThelium FT (HCT/P 361)+ SOC (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT (HCT/P 361)

INTERVENTIONS:
Other: NeoThelium FT (HCT/P 361) — NeoThelium FT is a dehydrated wound covering derived from donated human placental tissue.

SUMMARY:
This is a prospective case series evaluating the efficacy and safety of NeoThelium FT Amnion Skin Graft in the Mangement of Venous Leg Ulcers

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will begin SOC plus NeoThelium FT weekly applications. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of venous leg ulcer or venous insufficiency with a lower extremity wound
3. Subject has an venous leg ulcer without infection or clinically visible exposed bone
4. Index wound is a minimum of 1 cm2 and a maximum of 30 cm2 at first treatment visit
5. Adequate circulation if wound is location on the lower extremity demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to informed consent OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to the first treatment visit.
6. Venous Leg Ulcer is being treated with compression therapy for 7 days prior to treatment visit 1
7. Index wound is free of necrotic debris prior to NeoThelium FT application
8. Female subjects of childbearing potential having a negative pregnancy test prior to the first treatment visit
9. Wound free of clinical signs/symptoms of infection (no purulent discharge or cellulitis) post-debridement during screening and prior to the first treatment visit.
10. Subject is able and willing to follow the protocol requirements
11. Subject had signed informed consent
12. If 2 or more wounds are present, the wounds must be separated by at least 2 cm

Exclusion Criteria:

1. Subject is unable to comply with protocol treatment
2. Presence of infection prior to screening.
3. Multiple VLUs on the same leg with < 2 cm separation from the target ulcer.
4. Subject has comorbid conditions that may compromise subject safety or wound healing in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders
5. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound.
6. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
7. Known contraindications or hypersensitivity to amniotic membrane products or components of NeoThelium FT.
8. Concurrent participation in alternative clinical trial that involves investigational drug or HCT/P interfering with wound treatment and/or healing.
9. Subject is pregnant or breastfeeding
10. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to the first treatment visit; or anticipated use of the above during the course of the study
11. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to enrollment
12. Index ulcer suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using manual measurement utilizing a ruler and physical examination.
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up
Time to Closure | 1-12 weeks
  Average number of grafts and/or weeks used to achieve wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, Study Chair — SygNola, LLC
Locations (2):
- United States (2):
  - MedCentris of Metairie, Metairie, Louisiana
  - MedCentris of Slidell, Slidell, Louisiana

IPD SHARING:
Plan to Share IPD: No